CLINICAL TRIAL: NCT00331656
Title: Non-Invasive Positive Pressure Mask Ventilation vs Extrathoracic Biphasic Cuirass Ventilation in Patients With Acute Respiratory Failure: A Randomized Prospective Study.
Brief Title: Comparative Study of Non-Invasive Mask Ventilation vs Cuirass Ventilation in Patients With Acute Respiratory Failure.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NIVCOMPARE-HMO-CTIL
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2006-05

CONDITIONS: Respiratory Insufficiency; Chronic Obstructive Pulmonary Disease; Pneumonia; Pulmonary Edema; Neuromuscular Diseases
Keywords: noninvasive; positive; cuirass; ventilation; respiratory; failure
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive; Pneumonia; Pulmonary Edema; Neuromuscular Diseases; Respiratory Aspiration

INTERVENTIONS:
Device: Non-invasive positive pressure mask ventilators
Device: Extrathoracic biphasic cuirass ventilator (RTX, Hayek)

SUMMARY:
Non-invasive ventilation has become increasingly important in the management of patients with acute respiratory failure. One of its major goals is to prevent the need for invasive ventilation, which is associated with numerous complications. This study compares the usefulness and safety of two noninvasive techniques which are used in Medical practice: Noninvasive positive pressure ventilation using a face mask and extrathoracic biphasic ventilation using a cuirass. Each of these techniques has advantages and disadvantages and both may not suit all patients. It is therefore important to compare the two in terms of effectiveness in preventing invasive ventilation and their side effects profile, so that we can improve our understanding and expertise in the treatment of patients in respiratory failure.

DETAILED DESCRIPTION:
Non-invasive ventilation is becoming a frequent and important treatment option for patients with acute respiratory failure, in order to avoid endotracheal intubation and associated complications. Non-invasive techniques include positive pressure mask ventilation, negative (iron lung) ventilation and extrathoracic biphasic cuirass ventilation. However, large, prospective randomized trials comparing these techniques are lacking.

This prospective, randomized study will compare the effectiveness and side effects of non-invasive positive pressure mask ventilation vs extrathoracic biphasic cuirass ventilation in patients with acute respiratory failure.

Methods: Medical patients with acute respiratory failure caused by different etiologies, not requiring immediate endotracheal intubation, will be randomized to receive either positive pressure via face mask or extrathoracic biphasic ventilation via cuirass. Clinical response and/or the need for intubation and mechanical ventilation will be assessed throughout the study. Cross-over to the alternative mode will be provided in case of intolerance or lack of response.

Study endpoints: Need for endotracheal intubation, ICU and hospital mortality, length of ventilation, length of ICU and hospital stay and complication rates using the two modes.

Importance & implications: No studies have yet compared these two modes of noninvasive ventilation in acute respiratory failure. This study can improve our understanding and evidence based knowledge in the treatment of patients with acute respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

Medical patients with acute respiratory failure caused by different etiologies:

COPD exacerbation, cardiogenic pulmonary edema, pneumonia, ARDS and neuromuscular disorders patients admitted to the Medical Intensive Care Unit

Exclusion Criteria:

Patients or family members who refuse consent for the study, Patients requiring endotracheal intubation, Post-operative patients, Patients who require sedation, Patients who are unconscious or uncooperative, Patients with acute severe asthma, Patients with massive or submassive pulmonary embolism, Patients in shock of any etiology who are hemodynamically unstable, Patients with upper airway obstruction, Patients with upper GI bleeding or epistaxis, Facial deformity or trauma, Patients who are unable to maintain a patent airway, Pregnancy, Patients under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Need for endotracheal intubation
ICU and hospital mortality using the two modes

SECONDARY OUTCOMES:
Length of ventilation
Length of ICU and hospital stay
Complication rates using the two modes.

CONTACTS AND LOCATIONS:
Overall Officials: Sigal Sviri, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Corrado A, Confalonieri M, Marchese S, Mollica C, Villella G, Gorini M, Della Porta R. Iron lung vs mask ventilation in the treatment of acute on chronic respiratory failure in COPD patients: a multicenter study. Chest. 2002 Jan;121(1):189-95. doi: 10.1378/chest.121.1.189. PMID 11796450
- [Background] Gorini M, Ginanni R, Villella G, Tozzi D, Augustynen A, Corrado A. Non-invasive negative and positive pressure ventilation in the treatment of acute on chronic respiratory failure. Intensive Care Med. 2004 May;30(5):875-81. doi: 10.1007/s00134-003-2145-9. Epub 2004 Jan 21. PMID 14735237
- [Background] Todisco T, Baglioni S, Eslami A, Scoscia E, Todisco C, Bruni L, Dottorini M. Treatment of acute exacerbations of chronic respiratory failure: integrated use of negative pressure ventilation and noninvasive positive pressure ventilation. Chest. 2004 Jun;125(6):2217-23. doi: 10.1378/chest.125.6.2217. PMID 15189944